CLINICAL TRIAL: NCT04625361
Title: A Single Center, Randomized, Double-Blind, Placebo-Controlled Study of Single/Multiple Ascending Doses to Evaluate the Safety, Tolerability, Pharmacokinetics, and Single Center, Randomized, Double-Blind, Two Periods, Crossover, Food Effect Study of HEC122505MsOH Tablets in Healthy Chinese Subjects
Brief Title: Single and Multiple Dose Safety, Tolerability, PK and Food Effect Study of HEC122505MsOH Tablets in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC122505-P-01/CRC-C2017
Record Dates: First submitted 2020-11-09; First posted 2020-11-12 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Single dose of HEC122505MsOH Tablets（pilot trial arm） (Experimental): Healthy subjects receive single dose of tablets HEC122505MsOH
  Interventions: Drug: HEC122505MsOH
- Single dose of HEC122505MsOH Tablets（Part 1， Cohort 1） (Experimental): Healthy subjects receive single dose of HEC122505MsOH or matching placebo
  Interventions: Drug: HEC122505MsOH
- Single dose of HEC122505MsOH Tablets（Part 1， Cohort 2） (Experimental): Healthy subjects receive single dose of HEC122505MsOH tablets or matching placebo
  Interventions: Drug: HEC122505MsOH
- Single dose of HEC122505MsOH Tablets（Part 1， Cohort 3,Fed/Fasting） (Experimental): Following an overnight fast of at least 10 hours, a single dose of HEC585 will be administered on 2 separate occasions (fasting and after meal) in a randomized crossover fashion with different food restrictions.
  Interventions: Drug: HEC122505MsOH
- Single dose of HEC122505MsOH Tablets（Part 1， Cohort 4） (Experimental): Healthy subjects receive single dose of HEC122505MsOH tablets or matching placebo
  Interventions: Drug: HEC122505MsOH
- Single dose of HEC122505MsOH Tablets（Part 1，Cohort 5） (Experimental): Healthy subjects receive single dose of HEC122505MsOH tablets or matching placebo
  Interventions: Drug: HEC122505MsOH
- Single dose of HEC122505MsOH Tablets（Part 1， Cohort 6） (Experimental): Healthy subjects receive single dose of HEC122505MsOH tablets or matching placebo
  Interventions: Drug: HEC122505MsOH
- Multiple doses of HEC122505MsOH Tablets（Part 2， Cohort 1） (Experimental): Healthy subjects receive multiple doses of HEC122505MsOH tablets or matching placebo
  Interventions: Drug: HEC122505MsOH
- Multiple doses of HEC122505MsOH Tablets（Part 2， Cohort 2） (Experimental): Healthy subjects receive multiple doses of HEC122505MsOH tablets or matching placebo
  Interventions: Drug: HEC122505MsOH
- Multiple doses of HEC122505MsOH Tablets（Part 2， Cohort 3） (Experimental): Healthy subjects receive multiple doses of HEC122505MsOH tablets or matching placebo
  Interventions: Drug: HEC122505MsOH

INTERVENTIONS:
Drug: HEC122505MsOH — Part2：Mulltiple doses once daily, up to 8 days

SUMMARY:
The Safety, Tolerability, Pharmacokinetic and Food Effect Study of HEC122505MsOH Tablets in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are willing and are able to provide a written informed consent to participate in the study.
2. Without Plann for pregnancy or pregnant within 3 months after enrollment throughout the trial.
3. Subjects aged between 18 and 45 (both inclusive) years old.
4. Healthy volunteers has a body weight ≥50 kg (for male) or ≥ 45kg (for female) and body mass index ≥18 and ≤28 kg/m2 at screening.
5. Subjects, who are healthy, as having no clinically significant abnormalities in vital signs, physical examination, clinical laboratory test results, Chest X-ray and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

1. Subjects with a positive serology for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies and/or TP antibodies at screening.
2. Patients with the following diseases of clinical significance, including but not limited to those with gastrointestinal, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental, or cardiovascular and cerebrovascular diseases.
3. nown allergic reactions or hypersensitivity to any excipient of the drug formulation(s)， anaphylaxis physique.
4. Use of any prescription or non-prescription medications within 14 days prior to initial dosing，Use of any drugs that inhibit or induce liver metabolism within 28 days before the first dose, or use of any of the following drugs within 28 days before the first dose: monoamine oxidase inhibitors, opioids, serotonergic drugs, sympathetic nerves Drugs, breast cancer resistance protein substrates, dopaminergic antagonists, etc.
5. Consume foods or beverages containing caffeine, xanthine, alcohol, and grapefruit within 48 hours prior to initial dosing.
6. Positive results from urine drug screen test.
7. History of alcoholism or drink regularly within 3 months prior to the study (defined as Alcohol consumption of > 21 units/week), or positive results from alcohol breath test.
8. Regular smoking of more than 10 cigarettes per day within 3 months before administration of study drug, or inability to refrain from smoking during the course of the study.
9. Donate blood or lose blood 400 mL or more within 1 month prior to initial dosing.
10. Subjects who plan to receive or have had organ transplants.
11. Females who are lactating/breastfeeding, or positive result from pregnancy test for women of child-bearing potential.
12. Subjects who participated in another clinical trial within 3 months prior to initial dosing.
13. Any other condition with in the opinion of the investigator would render the patient unsuitable for inclusion in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

PRIMARY OUTCOMES:
The Number of Adverse Events (AEs) | Part 1：up to 6 days; Part 2: up to 13 days.
  To investigate the safety and tolerability of HEC122505MsOH by assessment of AEs (non-serious and serious) following administration of oral HEC122505MsOH tablets

SECONDARY OUTCOMES:
Cmax | up to 120 hours
  Maximum Plasma Concentration(Cmax)
AUC | up to 120 hours
  Area Under the Curve(AUC)
Tmax Tmax | up to 120 hours
  Maximum Peak Time(Tmax)
t½ | up to 120 hours
  Elimination Half-life(t½)
MRT | up to 120 hours
  Mean Residence Time(MRT)
CL/F | up to 120 hours
  Apparent Clearance(CL/F)
Vz/F | up to 120 hours
  Apparent Volume of Distribution(Vz/F)
Kel | up to 120 hours
  Elimination Rate Constant(Kel)

OTHER OUTCOMES:
MAO-B | up to 120 hours
  Monoamine Oxidase B（MAO-B）
MAO-A | up to 120 hours
  Monoamine Oxidase A（MAO-A）

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No